CLINICAL TRIAL: NCT01907373
Title: Effect of Probenecid on Pharmacokinetics, and Tolerability of Olmesartan in Healthy Chinese Volunteers
Brief Title: Drug Interaction Study of Olmesartan in Healthy Chinese Volunteers
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Central South University (Other)
Responsible Party: Principal Investigator, Kunyan Li, Center of New Drug Clinical Trial, Hunan Provincial Tumor Hospital (The Affiliated Tumor Hospital of Xiangya Medical School of Central South University), Central South University
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 200704
Record Dates: First submitted 2013-07-22; First posted 2013-07-25 (Estimated); Last update posted 2013-07-25 (Estimated); Status verified 2013-07

CONDITIONS: Drug Interaction of Olmesartan in Healthy Chinese Volunteers
Keywords: olmesartan; probenecid; pharmacokinetics; tolerability
MeSH Terms: interventions — Olmesartan Medoxomil

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- olmesartan medoxomil, PK of olmesartan (Active Comparator): drug: olmesartan medoxomil; dosage form: oral tablet; dosage: 20mg/time; frequency: once a day; duration: 4 days
  Interventions: Drug: olmesartan medoxomil
- olmesartan medoxomil+probenecid, PK of olmesartan (Experimental): drug1: olmesartan medoxomil; dosage form: oral tablet; dosage: 20mg/time; frequency: once a day; duration: 4 days; drug2: probenecid; dosage form: oral tablet; dosage: 500mg/time; frequency: 2 times/day; duration: 1 day
  Interventions: Drug: olmesartan medoxomil+probenecid

INTERVENTIONS:
Drug: olmesartan medoxomil
  Other Names: BENICAR; CS-866
  Arms: olmesartan medoxomil, PK of olmesartan
Drug: olmesartan medoxomil+probenecid
  Arms: olmesartan medoxomil+probenecid, PK of olmesartan

SUMMARY:
Hypertension and hyperuricaemia are widespread conditions. There is significant overlap between the two conditions. Serum uric acid (SUA) is currently recognized as a risk factor for cardiovascular disease. Thus, at some point in their therapy, hypertensive patients with hyperuricaemia are likely to require concurrent treatment with anti-hypertensive and hypouricaemic agents. For this reason, it is important to determine whether there are any pharmacokinetic interactions resulting from the concomitant administration of such agents.Olmesartan is an angiotensin II receptor antagonist and effective and well tolerated in the treatment of arterial hypertension. Probenecid is a well-established hypouricaemic agent for the treatment of hyperuricaemia and gout.The goal of this study was to examine the impact of coadministration of probenecid on the pharmacokinetic parameters and tolerability of olmesartan in healthy volunteers.

DETAILED DESCRIPTION:
Probenecid is a well-established hypouricaemic agent for the treatment of hyperuricaemia and gout and is thought to act on urate transporter 1 (URAT1), a novel member of the organic anion transporter (OAT) family, thereby increasing uric acid excretion in the kidney by blocking urate reuptake, and then, resulting in a decrease of SUA.

Olmesartan is an angiotensin II receptor antagonist and effective and well tolerated in the treatment of arterial hypertension. Olmesartan is orally administered in the prodrug form, olmesartan medoxomil, which is converted to the pharmacologically-active compound olmesartan upon de-esterification by the enzyme arylesterase in the intestinal wall, portal blood, and liver. Olmesartan is excreted by hepatobiliary and renal systems without further metabolism, and its pharmacokinetic profile is not affected by age or gender. In addition, the pharmacokinetic and pharmacodynamic profile of olmesartan is favorable, both in terms of providing effective 24-hour blood pressure (BP) control with once-daily dosing, and in restricting the likelihood of pharmacokinetic interactions with other drugs. Studies in vitro show organic anion transporting polypeptide 1B1 (OATP1B1), OATP1B3, multidrug resistance-associated protein 2 (MRP 2), and breast cancer resistance protein (BCRP) are involved in hepatobiliary and renal transport of olmesartan. We know probenecid interferes with the kidneys' organic anion transporter (OAT). Will probenecid have effects on the pharmacokinetics of olmesartan thereby result in changes of antihypertensive effect and side effects of olmesartan? Until now, many clinical studies have shown olmesartan has no pharmacokinetic interactions with other drugs; moreover, there is no research about the interactions between olmesartan and probenecid. In this study, we assess the involvement of probenecid in the pharmacokinetics and tolerability of olmesartan.

ELIGIBILITY:
Inclusion Criteria:

* written informed consent obtained,
* age 18 to 40 years and a body mass index between 19 and 25 kg/m2;
* negative test results for HIV and hepatitis В and C non-smoking status and
* an unremarkable clinical history

Exclusion Criteria:

* has history or evidence of a renal, gastrointestinal, hepatic, or hematologic abnormality or
* any acute or chronic disease, or
* an allergy to any drugs

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 12 (Actual)
Dates: Start 2009-08; Primary Completion 2009-09 (Actual); Study Completion 2009-10 (Actual)

PRIMARY OUTCOMES:
pharmacokinetic parameters | 48 hours after last administration of olmesartan medoxomil
  pharmacokinetic parameters:AUC0-48, AUC0→∞ and Css-av , tmax, t1/2, Css-max, and Css-min

SECONDARY OUTCOMES:
vital signs | at baseline (0) and at 1, 2, 3, 6, 12, 36, and 48 hours after last dosage of olmesartan medoxomil administration
  vital signs: blood pressure, heart rate, and respiratory rate

OTHER OUTCOMES:
Laboratory tests | at baseline and after completion of the study during 48 hours
  biochemistry and hematology test, routine urine test
electrocardiography | at baseline and after completion of the study during 48 hours

CONTACTS AND LOCATIONS:
Overall Officials: Kunyan Li, phD, Principal Investigator — Center of New Drug Clinical Trial, Hunan Provincial Tumor Hospital (The Affiliated Tumor Hospital of Xiangya Medical School of Central South University); Nong Yang, MS, Study Director — Center of New Drug Clinical Trial, Hunan Provincial Tumor Hospital (The Affiliated Tumor Hospital of Xiangya Medical School of Central South University)
Locations (1):
- Center of New Drug Clinical Trial, Hunan Provincial Tumor Hospital (The Affiliated Tumor Hospital of Xiangya Medical School of Central South University), Changsha, Hunan, China

REFERENCES:
- [Derived] Li KY, Qiu Y, Jiang Y, Luo CH, Lin XP, Wang J, Yang N. Effect of probenecid on pharmacokinetics and tolerability of olmesartan in healthy chinese volunteers. Curr Ther Res Clin Exp. 2014 Jan 9;76:7-10. doi: 10.1016/j.curtheres.2013.11.004. eCollection 2014 Dec. PMID 25067982